CLINICAL TRIAL: NCT00024453
Title: The Use of Teicoplanin in the Treatment of Septicaemia Caused by Coagulase-Negative Staphylococci - A Randomized Study Comparing Bolus Injection With Infused and/or Line-Locked Teicoplanin
Brief Title: Teicoplanin in Treating Septicemia in Patients Who Are Receiving Chemotherapy Through a Central Venous Catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CCLG-SC-1999-01; CDR0000068944 (Registry Identifier: PDQ (Physician Data Query)); EU-20124
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2009-06

CONDITIONS: Infection
Keywords: infection
MeSH Terms: conditions — Infections | interventions — Teicoplanin

INTERVENTIONS:
Biological: teicoplanin

SUMMARY:
RATIONALE: Giving the antibiotic teicoplanin by infusion and allowing bacteria to be exposed to the antibiotic for a longer period of time may be effective in preventing or controlling septicemia.

PURPOSE: Randomized clinical trial to compare two different methods of giving teicoplanin in treating septicemia in patients who are receiving chemotherapy through a central venous catheter.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response and cure rate of coagulase-negative staphylococcal septicemia in patients receiving chemotherapy through a central venous catheter treated with 2 different schedules of teicoplanin.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center and number of central venous catheter lumens (1 vs 2). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive teicoplanin IV bolus every 12 hours for 3 doses and then once daily for 5 doses (total of 7 days).
* Arm II: Patients receive teicoplanin IV over 2 hours and/or by antibiotic lock every 12 hours for 3 doses and then once daily for 5 doses (total of 7 days).

PROJECTED ACCRUAL: Approximately 490-1,360 patients will be accrued for this study within 2.2-6.2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Suspected septicemia caused by coagulase-negative staphylococci
* Single or double lumen (no triple lumen) central venous catheter (CVC) (including subcutaneous ports) that can be flushed and aspirated

  * Expected to remain in situ for at least 8 weeks
* No coagulase-negative septicemia associated with existing CVC within the past 12 weeks
* Receiving chemotherapy for neoplastic condition, aplastic anemia, Fanconi's anemia, Langerhans' cell histiocytosis, or myelodysplasia

PATIENT CHARACTERISTICS:

Age:

* 2 months and over

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Creatinine clearance at least 60 mL/min

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1360 (Estimated)
Dates: Start 1999-02; Primary Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Pizer, MD, Study Chair — Royal Liverpool Children's Hospital, Alder Hey
Locations (21):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Bristol Royal Hospital for Children, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Saint Bartholomew's Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - University College of London Hospitals, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Newcastle Upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland